CLINICAL TRIAL: NCT01965041
Title: Use Of Intravitreal Aflibercept Injections In The Treatment Of Adult-Onset Vitelliform Detachments Associated With Pattern Dystrophy
Brief Title: Intravitreal Aflibercept Injections In The Treatment Of Pattern Dystrophy
Acronym: AVA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The AVA Study
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Pattern Dystrophy of Macula
Keywords: AVA Study
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eyelea, ophthalmic exam, photgraphy (Experimental): 2.0 mg intravitreal aflibercept injection is formulated as a sterile liquid to a final concentration of 40 mg/mL aflibercept in 5% sucrose, 10 mM sodium phosphate pH 6.3, 0.03% polysorbate 20, and 40 mM NaCl
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — 2.0 mg intravitreal aflibercept injection is formulated as a sterile liquid to a final concentration of 40 mg/mL aflibercept in 5% sucrose, 10 mM sodium phosphate pH 6.3, 0.03% polysorbate 20, and 40 mM NaClvs. placebo
  Other Names: eylea

SUMMARY:
Adult-onset vitelliform detachments associated with pattern dystrophy is a genetic disorder that carries visual implications that most commonly affect the macula (area in the eye near the retina that is essential for sharp central vision). Adult onset vitelliform detachments have an accumulation of material on the outer retina. Over time, the abnormal accumulation of this material can damage cells that are critical for clear central vision. As a result, people with this disorder often lose their central vision, and their eyesight may become blurry or distorted.

DETAILED DESCRIPTION:
Subretinal fluid is thought to play a role in the formation of vitelliform detachments, which are associated with progressive vision loss. Fluid in the subretinal space disrupts the physical apposition between photoreceptor outer segments and retinal pigment epithelial cells, which may in turn hinder the phagocytosis of shed photoreceptor outer segments. Material derived from the unphagocytized outer segments may accumulate in the subretinal space to form vitelliform lesions, resulting in a persistent detachment. Anti-VEGF therapy in the form of intravitreal aflibercept injections may be useful in controlling or eliminating subretinal fluid, thus promoting contact between photoreceptor outer segments and the retinal pigment epithelium. Vitelliform detachments may resolve subsequent to the removal of subretinal fluid and restoration of contact-dependent mechanisms of photoreceptor outer segment recycling.

ELIGIBILITY:
Inclusion Criteria:A patient must meet the following criteria to be eligible for inclusion in the study:

1. Presence of adult onset vitelliform detachment associated with pattern dystrophy of at least one year duration 2. Treatment naive 3. Age >50 years old 4. Willing and able to comply with clinic visits and study-related procedures 5. Provide signed informed consent

-

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Previous treatment of adult onset vitelliform detachment associated with pattern dystrophy
2. Presence of any substantial ocular disease that may compromise or confound interpretation of the data
3. Active intraocular inflammation
4. Patients allergic to fluorescein, povidone iodine (Betadine) or aflibercept
5. Patients on systemic anti-VEGF agents within 3 months of study enrollment
6. Participation in a study of an investigational drug or device within 30 days prior to potential enrollment into the study
7. Pregnant or breast-feeding women
8. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

   * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
• The incidence and severity of systemic and ocular adverse events. | 0 - 6 months

SECONDARY OUTCOMES:
• Anatomic reduction or resolution of vitelliform as determined by change on OCT, FA, fundus photos, and autofluoresence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, M.D., Principal Investigator — Northshore Long Island Jewish Healthcare Systems
Locations (1):
- Ns/Lij Meeth, New York, New York, United States